

# UNIVERSITY OF PENNSYLVANIA RESEARCH SUBJECT INFORMED CONSENT FORM AND HIPAA AUTHORIZATION

**Protocol Title:** The COMET-PCOS trial- Comparing the effects of

Oral Contraceptive Pills versus Metformin in the medical management of overweight/obese women

with Polycystic Ovary

**Principal** Anuja Dokras, MD, PhD

**Investigator** 3701 Market Street, Suite 800

University of Philadelphia, PA 19104

**Pennsylvania**: 215-615-0085

Principal Monica Mainigi, MD

Investigator The Children's Hospital of Philadelphia

**Children's** 34th Street and Civic Center Blvd.

Hospital of Philadelphia, PA 19104

**Philadelphia:** 215-662-2972

**Emergency** Fellow On Call **Contact:** 215-662-6100

# Why am I being asked to volunteer?

You are being invited to participate in a research study because you have Polycystic Ovary Syndrome (PCOS) and are overweight. Your participation is voluntary which means you can choose whether or not you want to participate. If you choose not to participate, there will be no loss of benefits to which you are otherwise entitled. Before you can make your decision, you will need to know what the study is about, the possible risks and benefits of being in this study, and what you will have to do in this study. The research team is going to talk to you about the research study, and they will give you this consent form to read. You may also decide to discuss it with your family, friends, or family doctor. You may find some of the medical language difficult to understand. Please ask the investigator and/or the research team about this form. If you decide to participate, you will be asked to sign this form. Your doctor may be an investigator in this research study. As an investigator, your doctor is interested both in your clinical

welfare and in the conduct of this study. Before entering this study or at any time during the research, you may want to ask for a second opinion about your care from another doctor who is not an investigator in this study. You do not have to participate in any research study offered by your doctor.

#### What is the purpose of this research study?

This research study is being conducted to determine the if there is an effect on Metabolic Syndrome (MetS) in overweight/obese women with PCOS when Oral Contraceptive Pills (OCP) are given in combination with Metformin. Metabolic Syndrome is the name for a group of risk factors that raises your risk for heart disease and other health problems, such as diabetes and stroke. Currently, there are no clear recommendations for the best and most comprehensive medical management of overweight/obese women with PCOS. The study hopes to uncover whether OCP and Metformin together affect the prevalence of MetS, thereby altering the risk profile for the development of diabetes and cardiovascular disease in women with PCOS.

## How long will I be in the study?

If you chose to participate in this study, your participation will last for 24 weeks (about 6 months). The study is being conducted at two medical centers, the University of Pennsylvania (UPenn) and Pennsylvania State University-Hershey Medical Center (PSU). The study hopes to recruit 240 women (approximately 120 women at each site). We will also be recruiting women with PCOS from Children's Hospital of Pennsylvania.

# What am I being asked to do?

If you chose to participate in this study, you must sign this consent form. You will be placed into one of three groups and asked to take the study medication for the duration of the study. You will either be assigned to one of three groups: 1) OCP + placebo pills, 2) Metformin + placebo pills, or 3) OCP + Metformin. Placebo pills are used as a control, meaning they do not contain any active medication (like a sugar pill). The use of a placebo will help the investigators understand what medications are having the greatest effect in the study. The OCP used for this study is 20mcg ethinyl estradiol/desogestrel 0.15mg. This is a low dose birth control pill that would have a lesser impact on lipids and insulin sensitivity as these lab values can sometimes be reported high in women with PCOS. Since the assigned treatment groups are randomized and blinded we do ask that you use a medically accepted non hormonal method of birth control (such as condoms) while you participate in the study.

You will be asked to come to the University of Pennsylvania for 6 study visits (a screening visit, randomization visit, 4 weeks, 8 weeks, 16 weeks and 24 weeks visit). The screening visit will determine if you are eligible to participate in the study. You may need to stop taking certain medications (wash-out) to participate in the study. A one-month wash-out period (6 month wash out in the case of injectable hormonal contraceptive) will be required for medications prior to screening (most common OCP and metformin). Some medications will be

prohibited during this study. Please discuss any medications you are taking with the study doctor. The study doctor will inform you of any medication that you need to stop.

If you are found to be eligible you will be randomized (assigned to a group by chance, like the flip of a coin) to one of the medication groups mentioned above. If you have not had a menstrual period for three months prior to the randomization visit, the study will induce menses through use of medication medroxyprogesterone acetate (MPA). Through-out the study, the research team will collect information about your medical and menstrual history, take your vital signs (height, weight, blood pressure and pulse) and draw your blood for screening and safety labs.

Please refer to the study schedule below for more information on the timing of the events to take place during each study visits and further details of specific events that will occur.

| Study Visit<br>Schedule | Screening<br>Visit | Randomization<br>Visit | 2 Week<br>PC | 4 Week<br>Visit | 8 Week<br>Visit | 12 Week<br>PC | 16 Week<br>Visit | 20 Week<br>PC | 24 Week<br>Visit | Safety<br>PC |
|---|---|---|---|---|---|---|---|---|---|---|
| Sign Informed<br>Consent | X | | | | | | | | | |
| Medical<br>Assessment | Х | | | | | | | | | |
| Review Menstrual history | Х | Х | Х | Х | Х | Х | Х | Х | X | Х |
| Urine Pregnancy test | Х | Х | | Х | Х | | Х | | X | |
| Vital Signs/<br>Biometrics | Х | Х | | Х | Х | | Х | | X | |
| Screening labs | X* | | | | | | | | | |
| Safety labs | X* | Х | | | | | Х | | Х | |
| Hirsutism (F-G) score | × | Х | | | | | | | × | |
| Acne assessment | | X | | | | | | | Х | |
| DXA | | Х | | | | | | | Х | |
| DNA Sample | | Х | | | | | | | | |
| Fasting blood draw | | Х | | | | | Х | | × | |
| Lifestyle<br>Modification<br>Counselling | | × | | | | | Х | | | |
| ASA24 | | | | | | Х | | | Х | |
| TVUS | X* | X | | | | | | | Х | |
| oGTT | | Х | | | | | | | Х | |
| Randomization | | X | | | | | | | | |
| PCOSQ/STAI/CE<br>S-D/FSDS-<br>R/FSFI | | X | | | | | | | Х | |
| Cognitive<br>Questionnaires | | Х | | | | | | | Х | |
| Review Adverse<br>Events | | | Х | Х | Х | Х | Х | Х | Х | Х |
| Review<br>Concomitant<br>Medications | Х | X | Х | Х | Х | Х | Х | Х | Х | Х |
| Dispense<br>Logs/Medications | | Х | | Х | Х | | Х | | | |
| Collect<br>Logs/Medications | | | | Х | Х | | Х | | X | |

<sup>\*</sup>As Needed

<u>Hirsutism Score:</u> Hirsutism is excessive hair that commonly appears in a male pattern in females and it is generally associated with hyperandrogenic PCOS. The Ferriman-Gallwey Hirsutism Score is used to evaluate hair growth in nine areas of the body.

<u>Urine Pregnancy Test:</u> A urine pregnancy test will be performed at all visits. If a positive result is found, you will be informed by the site staff of the positive result and offered resources regarding prenatal care or alternative options.

<u>Lifestyle Modification Counseling:</u> You will receive counseling about diet and exercise at the randomization and 4-month visit. The diet will be designed to reduce your calorie intake by 500 calories a day.

<u>ASA24:</u> The Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24). This 24-hour dietary recall captures detailed information about all foods, drinks, and supplements (including vitamins, minerals, herbals, and other dietary supplements) you consumed from midnight to midnight. You will be asked to complete this at 12 weeks and 24 weeks.

<u>Questionnaires (PCOSQ, STAI, CES-D, FSDS-R, FSFI):</u> The <u>PCOSQ</u> is self-administered questionnaire for measuring health-related quality of life in women with PCOS. The PCOSQ will be at randomization and the 24 weeks visit. The <u>STAI</u> (State-Trait Anxiety index) is a questionnaire for accessing trait anxiety and state anxiety. The STAI will be administered to subjects at Randomization and 24 week visit. The <u>CES-D</u> is a screening test for depressive symptoms. The CES-D will be administered to subjects at Randomization and 24 week visit. The <u>FSDS-R</u> (The Female Sexual Distress Scale-Revised) is a screening questionnaire for measuring sexually related personal distress in women with Female Sexual Dysfunction (FSD). The <u>FSFI</u> (Female Sexual Function Index) is a brief questionnaire measure of sexual function in women. It was developed for the specific purpose of assessing domains of sexual function (e.g. sexual arousal, orgasm, satisfaction, pain) in clinical trials.

<u>Transvaginal ultrasound:</u> a transvaginal ultrasound will be performed to look at your ovaries (the female reproductive organ where eggs are produced). This will occur at the screening (if needed), randomization visit and 24 weeks visit.

<u>DXA Scan:</u> a DXA scan will be performed to take a measure of your bone density.

<u>Oral Glucose Test (oGTT):</u> measures the body's ability to use a type of sugar, called glucose, that is the body's main source of energy. This will be performed at the randomization and 24 weeks visit. Prior to the test, you must fast overnight for 10-14 hours. You will receive an oral glucose solution and your blood will be sampled every 30 minutes for 2 hours. (An IV will be inserted if you desire to avoid multiple blood draws).

<u>Cognitive Testing</u>: test designed to measure an individual's cognitive (thinking, reasoning or remembering) function in a specific area, such as verbal reasoning, spatial awareness or mathematics. Audio recording of cognitive testing is optional. If you chose to be audio recorded- it will be deleted after transcription.

<u>Blood banking:</u> If you agree, your blood will be collected and stored in the repository and used for future research that has not yet been defined.

<u>Genetic testing:</u> If you agree, your blood will also be used to obtain a sample of your genetic material (DNA). We will use these samples for genetic research, which might teach us about health conditions that are passed on in families. The purpose of collecting your DNA and how it will be used is discussed further in this consent form. If you decide that you do not want your DNA collected, you will still be able to participate in this study

### What are the possible risks or discomforts?

Risk are addressed by using trained medical staff, close observation and contact with you throughout the study. The possible risk of participating in this study include:

<u>Blood Samples:</u> Possible side effects from blood drawing include feeling faint, inflammation of the vein, pain, bruising, or bleeding at the site of puncture. There is a slight possibility of infection at the site or draw. The blood testing performed outside of Penn will be conducted at the Children's Hospital of Pennsylvania (CHOP) Translational Core Lab (TCL), Michigan University, and National Institutes of Health.

<u>Oral Glucose Test:</u> Possible side effects from this test include anemia (lack of red blood cells), infection at the site of the IV, nausea, vomiting, allergic reaction, hypoglycemia (low blood sugar), as well as all the standard blood draw discomforts and risks.

<u>Transvaginal ultrasound:</u> Possible side effects include abdominal or pelvic discomfort.

<u>Reduced Calorie Diet:</u> Possible side effects include hunger, weakness, changes in your electrolytes (salts in your body), mood changes, depression, gall stone from rapid weight loss.

<u>Oral Contraceptive Pills:</u> Possible side effects include abdominal bloating, cramps, or pain, nausea, breast tenderness, mood changes, weight changes, headaches, breakthrough bleeding, blood clot, stoke, elevated blood pressure, gallbladder disease, swelling, irritated varicose vein, depression, migraine, absence of a cycle, breast changes, appetite changes, vomiting, fluid retention, temporary infertility, menstrual flow changes, spotting.

<u>Metformin:</u> The most common side effects of this drug are gastrointestinal symptoms (diarrhea, nausea, vomiting, abdominal bloating, flatulence, metallic taste in mouth and anorexia). There is a small risk of lactic acidosis (a medical condition when cells make lactic acid, from glucose, faster than the body can break it down).

Medroxyprogesterone acetate (MPA): Possible side effects include abnormal uterine bleeding (irregular, increase, decrease), change in menstrual flow, breakthrough bleeding, spotting, no menses, changes in cervical erosion and cervical secretions, breast pain or tenderness, nausea, cholestatic jaundice, swelling, generalized rash, acne, hair growth, hair loss, depression, insomnia, sleepiness, dizziness, headache, nervousness, hypersensitivity reactions, rash (allergic) with and without itching of skin, change in weight (increase or decrease), increased body temperature, fluid retention, fatigue, decreased glucose tolerance.

<u>DXA Scan:</u> Exposure to a small amount of x-ray radiation. Therefore, you will receive a radiation dose. This radiation dose is not necessary for your medical care and will occur only as a result of your participation in the study. At doses much higher than you will receive, radiation is known to increase the risk of developing cancer after many years. At the doses you will receive, it is very likely that you will see no effects at all.

<u>Questionnaires:</u> Some questions may make you feel embarrassed or uncomfortable. You do not have to answer any questions which make you uneasy.

Reproductive risks: Because of the effects of these drugs there could be serious harm to unborn children or children who are breast-feeding. These effects could also harm the mother. It is also possible that harmful side effects that are not yet known could happen to both the mother and unborn or breast-feeding child. If you are currently pregnant, it is important that you inform the investigator because you will not be able participate in the study. If you are able to become pregnant, you will be given a serum pregnancy test before entry into the study. Since we will not know which study participants have received an OCP, you are asked to use a medically accepted non hormonal method of birth control (such as condoms) while you participate in the study. You should not become pregnant while you are taking these drugs. If you do become pregnant, you must tell the investigator immediately and you will be discontinued from the study. Some information will be gathered from you regarding the pregnancy, including the completion of a transvaginal ultrasound. You will be referred to consult an obstetrician or maternal-fetal specialist.

#### Risks of Genetic Testing:

This research includes optional genetic testing. Even without your name or other identifiers, your genetic information is unique to you. The researchers believe the

chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information.

There can be a risk in knowing genetic information. New health information about inherited traits that might affect you or your blood relatives could be found during a research study. Even though your genes are unique, you share some of the same genes with your blood relatives. Although we are not able to know all of the risks from taking part in research on inherited traits, we believe that the risks to you and your family are very low, because your samples will be coded. Research results will not be returned to you or your doctor.

Very rarely health or genetic information could be misused by employers, insurance companies, and others. For example, it could make it harder for you to get or keep a job or insurance, or life insurance companies may charge a higher rate based on this information. We believe the chance these things will happen is very small, but we cannot make guarantees.

A federal law (Genetic Information Non-Discrimination Act, GINA) helps reduce the risk from health insurance or employment discrimination. The law does not include other types of misuse by life insurance or long term care insurance. If you want to learn more about GINA, you can find information about it on the internet or ask the study staff.

Loss of Confidentiality: There is a risk of loss of confidentiality if your information or your identity is obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your electronic data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

<u>Unforeseen Risk:</u> Since the study is investigational there may be risks that are unknown. If you experience any adverse reactions, please contact the study doctor/staff and seek medical help if necessary.

For this study we may need to contact you via email or test message to provide you information about scheduling, appointments notes, or to send you information about your participation in the study. Email and text communications are often not secure and may be seen by others as a result. For test messages, message and data rates may apply to you while enrolled. By signing below, you accept these risks and potential additional costs.

If you wish for us to use a different means to communicate with you during the course of this trial, please discuss this with the research team and alternative methods can be arranged. You can text "stop" to any text message to opt-out of the text messaging program.

## What if new information becomes available about the study?

During the course of this study, we may find more information that could be important to you. This includes information that, once learned, might cause you to change your mind about being in the study. We will notify you as soon as possible if such information becomes available.

# What are the possible benefits of the study?

You may benefit as a result of your participation in this study. You may experience improvements in symptoms associated with PCOS. There is, however, no guarantee that you will benefit from your participation in this study. It is possible that information from the use of these study drugs may help advance knowledge for development of more effective treatment of women with PCOS in the future. Result of this study may benefit others.

# What other choices do I have if I do not participate?

You do not have to participate in this study to receive treatment of your PCOS. You may receive standard of care through the University of Pennsylvania PCOS Center or Children's Hospital of Philadelphia.

## Will I be paid for being in this study?

For your time and inconvenience related to your participation in this study, you will be paid for the study visits you complete. You will be paid as follows:

Screening visit = \$50
Randomization visit = \$125
Week 4 visit = \$50
Week 8 visit = \$50
Week 16 visit = \$50
Week 24 visit = \$125

You may also be paid \$50 for any unscheduled study visit. We will pay you by using a Greenphire ClinCard which is a pre-paid debit card in which your payment will occur at the end of each visit you attend. After giving you the card at the screening visit, the card will be loaded with additional payments at every scheduled visit.

Please note: In order to be compensated for your participation in this study, you must provide your Social Security Number. Additionally, please note that the University of Pennsylvania is required to report to the IRS any cumulative payments for participation in research studies that exceed a total of \$600 in a calendar year.

#### Will I have to pay for anything?

There will be no charge to you for your participation in the study. The study drug, study-related procedures and study visits will be provided at no charge to you or your insurance. Please note any clinical procedure you have outside the study at the University of Pennsylvania will be your responsibility.

## What happens if I am injured from being in the study?

We will offer you the care needed to treat injuries directly resulting from taking part in this research. We may bill your insurance company or other third parties, if appropriate, for the costs of the care you get for the injury, but you may also be responsible for some of them.

There are no plans for the University of Pennsylvania to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

If you think you have been injured as a result of taking part in this research study, tell the person in charge of the research study as soon as possible. The researcher's name and phone number are listed in the consent form.

# When is the Study over? Can I leave the Study before it ends?

This study is expected to end after all participants have completed all visits, and all information has been collected. This study may also be stopped at any time

by your physician, the study Sponsor, or the Food and Drug Administration (FDA) without your consent because:

- The Primary Investigator feels it is necessary for your health or safety. Such an action would not require your consent, but you will be informed if such a decision is made and the reason for this decision.
- You have not followed study instructions.
- The Sponsor, the study Principal Investigator, or the Food and Drug Administration (FDA) has decided to stop the study.

If you decide to participate, you are free to leave the study at anytime. Withdrawal will not interfere with your future care.

# Who can see or use my information? How will my personal information be protected?

We will do our best to make sure that the personal information obtained during the course of this research study will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. The Institutional Review Board (IRB) at the University of Pennsylvania will have access to your records. If this study is being overseen by the Food and Drug Administration (FDA), they may review your research records. We will use study ID numbers to identify your data and specimens. The list that matches your name with your study ID number will be kept in a secured area in a locked filing cabinet or in a password-protected electronic document at University of Pennsylvania. This list will be kept indefinitely.

Your samples may be used to create products, including some that may be sold and/or make money for others. If this happens, there are no plan to tell you, or to pay you, or to give any compensation to you or your family.

## Will information about this study be available to the public?

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

## Future use of Data and/or Specimens

Your information and samples coded with your study ID number will be stored for future research purposes. Future researchers may receive information that could identify you. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information and samples only applies to the information and samples collected on this study. Your study ID number will be retained and shared with data/samples. Your information and samples

may be stored and used for future research purposes for an indefinite amount of time.

There are no plans to tell you about any specific research that will be done. Possible future research may include additional research on PCOS or metabolic syndrome. We may share your identifiable information and samples with other researchers.

We will not follow up with you to tell you about the specific research that will be done. We will not give you any results from these studies. It is possible that you may have chosen not to participate in these future research studies, had you been approached for participation.

There is a risk of breach of confidentiality (unintentional release of your information). We will do our best to make sure that this doesn't happen. However, we cannot guarantee total privacy. We will protect your confidentiality during storage and sharing by keeping the list which matches your name with your study ID number in a secured area in a locked filing cabinet or in a password-protected electronic document at University of Pennsylvania.

You will likely not directly benefit from future research with your information and samples. Research with your identifiable information and samples may help others by improving our understanding of health and disease, improving health care and making safer or more effective medical therapies, and developing new scientific knowledge.

If you have questions about the storage of your information and samples or have changed your mind about use of your samples, you should contact Dr. Dokras in writing at the address on page 1 of this form. Once the samples have left the University of Pennsylvania or have been completely used there is no way to have them returned or withdrawn for testing. You will not be able to withdraw your permission for future use at that time. Any analysis or test results already performed will be kept. Information that has already been used or shared with others will be retained.

# Electronic Medical Record and Release of Study Related Information

#### What is an Electronic Medical Record?

An Electronic Medical Record (EMR) is an electronic version of your medical chart within a health system. An EMR is simply a computerized version of a paper medical record.

If you have never received care within Penn Medicine and are participating in a University of Pennsylvania research study that uses Penn Medicine healthcare related services, an EMR will be created for you for the purpose of maintaining any information produced from your participation. The creation of this EMR is a requirement of your participation in this study. In order to create your EMR, the study team will need to obtain basic information about you that would be similar

to the information you would provide the first time you visit a hospital or medical facility (i.e. your name, the name of your primary doctor, the type of insurance you have). If you have been a patient at Penn Medicine in the past, information from your research participation will be added to your existing medical record.

#### What may be placed in the EMR?

Information related to your participation in the research (e.g., laboratory tests, notes from your physician, imaging studies, and clinical procedures, etc.) will be placed in your EMR maintained by Penn Medicine.

Once placed in your EMR your information may be accessible to appropriate Penn Medicine workforce members that are not part of the research team. Information within your EMR may also be shared with others who are determined by Penn Medicine to be appropriate to have access to your EMR (e.g. Health Insurance Company, disability provider, etc.).

Penn Medicine also participates in automated information sharing through Health Information Exchanges (HIEs). HIEs securely share parts of your electronic health record, including research information, with other healthcare organizations involved in your care. This information is shared to improve the quality, safety and efficiency of your healthcare. To request that your health information not be shared through HIEs, please call 215-662-4484.

# Will I, as a subject, have access to research related information within the EMR?

The 21st Century Cures Act requires healthcare institutions to allow patients increased access to their electronic medical record. As part of your participation in this research, you will have access to research related information within your EMR through Penn Medicine's patient portal – called MyPennMedicine (MPM).

Some information specific to this clinical research study may be shared with you in a delayed manner, shared with you at the end of the study, or not shared with you. Not sharing or delaying certain research information within your EMR may be necessary to protect the integrity of the trial results or for other reasons.

# Will I receive the results of research testing that may be relevant to my health?

Many of tests done in research studies are only for research and have no clear impact on your healthcare. Research results for this study will not be returned to you because they would not be relevant to your healthcare.

# Who can I call with questions, complaints or if I'm concerned about my rights as a research subject?

If you have questions, concerns or complaints regarding your participation in this research study or if you have any questions about your rights as a research subject, you should speak with the Principal Investigator listed on page one of this form. If a member of the research team cannot be reached or you want to

talk to someone other than those working on the study, you may contact the Office of Regulatory Affairs with any question, concerns or complaints at the University of Pennsylvania by calling (215) 898-2614.

If you are a CHOP patient/subject and have questions about your rights or if you have a complaint, you can call the CHOP Office of Research Compliance at 215-590-2830.

# What information about me may be collected, used or shared with others?

During your participation in this research study, the study investigator and study staff will collect personal health information about you (for example, medical histories and result of any tests, examinations or procedures you undergo while in the study) and record it on study documents. The study investigator will keep this personnel health information in your study related records. In addition, the study doctor may obtain, and include in your records, information regarding your past, present and/or future physical or mental health and/or condition. Your study investigator may ask you to sign a separate authorization to obtain some or all of your medical records from your study doctor. Your study records may include other personal information (such as name, social security number, medical record numbers, date of birth, address, telephone number, and email address) which could identify you. Health information that could identify you is call "Protected Health Information" (or PHI).

Under federal law (the "Privacy Rule"), your PHI that is created or obtained during this research study cannot be "used" to conduct the research or "disclosed" (given to anyone) for research purposes without your permission. This permission is called an "Authorization". Therefore, you may not participate in this study unless you give your permission to use and disclose you PHI by signing this Authorization. By signing, you are agreeing to allow the study investigator and staff to use you PHI to conduct this study.

# Why is my information being used?

Your information is used by the research team to contact you during the study. Your information and results of tests and procedures are used to:

- do the research
- oversee the research
- to see if the research was done right
- to evaluate and manage research functions.

## Where may my information be stored?

Information related to your participation in clinical research will be contained in a clinical trial management system (CTMS). A clinical trial management system (CTMS) is used to register your information as a participant in a study. This allows for your research data to be entered and stored for the purposes of study operational and financial applications and other activities required as part of the conduct of the research. Once placed in the CTMS your information may be

accessible to other authorized personnel at Penn Medicine that support research operations. Your information may be held in other research databases.

#### Who may use and share information about me?

The following individuals may use or share your information for this research study:

- The investigator for the study and the study team
- Other authorized personnel at Penn, including offices that support research operations
- The investigator for the study at PSU- Hershey Medical Center
- The investigator for the study at CHOP and the Children's Hospital of Pennsylvania (CHOP) Translational Core Lab (TCL)
- Other research personnel with access to the databases for research and/or study coordination and as otherwise approved by the IRB

# Who, outside of the School of Medicine, might receive my information?

List all names or all classes of persons involved in the research at Penn, e.g.,

- Greenphire ClinCard
- Those working under the direction of the investigator for the study, (e.g. under subcontracts).
- All research centers participating in the study, even if they are not part of the School of Medicine
- The funding sponsor and organizations supporting the sponsor

#### Oversight organizations

- The Food and Drug Administration
- The Office of Human Research Protections
- The study data and safety monitoring board
- Michigan University
- National Institutes of Health.

Once your personal health information is disclosed to others outside the School of Medicine, it may no longer be covered by federal privacy protection regulations.

The Principal Investigator or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to University of Pennsylvania procedures developed to protect your privacy.

# How long may the School of Medicine use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study does not expire.

Your information may be held in a research database. However, the School of Medicine may not re-use or re-disclose information collected in this study for a purpose other than this study unless:

- You have given written authorization
- The University of Pennsylvania's Institutional Review Board grants permission
- As permitted by law

# Can I change my mind about giving permission for use of my information?

Yes. You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the investigator for the study (listed on the top of this form). If you withdraw your permission, you will not be able to stay in this study.

If you withdraw your permission, we will stop collecting health information about you for this study; we may continue to use and share your health information that we already have if it is necessary for safety and scientific soundness of the research study; and we will not be able to take back information that has already been used or shared with others.

# What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study.

You will be given a copy of this Research Subject HIPAA Authorization describing your confidentiality and privacy rights for this study.

By signing this document, you are permitting the School of Medicine to use and disclose personal health information collected about you for research purposes as described above.

#### **Decisions**

#### Optional DNA, Blood Collection:

As part of this study, we are obtaining, prior to you starting medication, a sample of your blood for DNA testing and for measure of other substances in the blood. If you agree, the researchers would like to use your DNA to identify certain sequences of key genes (called polymorphisms) that may predict a response to the medications used in this trial. If genes are identified, which are related to the response to the treatment, the sample may also be used in the development of diagnostic or prognostic tests to identify those who will or who will not respond to these medications. We also may use this DNA to identify genes that cause PCOS. Additionally, we are banking part of your blood that does not contain cells to eventually study proteins that are determined by these genes. There is no normal or abnormal result produced by the DNA or blood tests, and the researchers will not use the DNA to try to see if you have any genetic diseases or conditions. The testing of DNA may provide additional information that will be helpful in understanding the medications used in this trial and the effects on PCOS, but it is unlikely that these studies will have a direct benefit to you. The results of these tests will not have an effect on your care. Neither your doctor nor you will receive results of these tests, and the results will not be put in your medical records.

If you agree to allow your DNA sample to be collected at the randomization visit. it will be stored in a secure laboratory at the study site. You are free to change your mind regarding the use of your sample. If you no longer want your DNA or blood to be used for testing, you should contact Dr. Dokras in writing at the address on page 1 of this form. Your DNA and blood sample will be destroyed at that time of withdrawal. If you consent to the collection of your DNA, it will be kept indefinitely or until the sample is used completely by the staff and collaborators of this study.

You should initial below to indicate your preference for the collection of your DNA sample:

#### **Optional Consent:**

| I agree to have an optional collection of blood which can be stored in the repository and used for future research that has not yet been defined. YES NO | |
|---|---|
| I agree to have an optional collection of blood for DNA testing which can stored in the repository and used for future research that has not yet beer defined. | |
| YES NO | |
| I agree to have an optional audio recording done during my cognitive test<br>help assess accuracy of my answers and standardization of the test<br>environment. | ing to |
| YES NO | |
| Version 9.0 –March 1, 2023 | 16 of 1 |

IRB Approval From: 05-16-2023 To: 05-15-2024

When you sign this form, you are agreeing to take part in this research study. This means that you have read the consent form, your questions have been answered, and you have decided to volunteer. Your signature also means that you are permitting the University of Pennsylvania to use your personal health information collected about you for research purposes within our institution. You are also allowing the University of Pennsylvania to disclose that personal health information to outside organizations or people involved with the operations of this study.

| A copy of this consent form wi | Il be given to you. | |
|--------------------------------|-------------------------|------|
| Name of Subject (Please Prin | t) Signature of Subject | Date |
| Name of Person Obtaining | Signature | Date |